CLINICAL TRIAL: NCT02594709
Title: Observational Study on Multisession Radiosurgery for Optic Nerve Sheath Meningiomas
Brief Title: Multisession Radiosurgery for Optic Nerve Sheath Meningiomas
Acronym: ONSMsmSRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRON-SM
Record Dates: First submitted 2015-10-15; First posted 2015-11-03 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Optic Nerve Sheath Tumors, Benign
MeSH Terms: conditions — Optic Nerve Neoplasms

STUDY DESIGN:
Intervention Model Description: Radiosurgery
Oversight: Data Monitoring Committee: No

ARMS (1):
- ONSM Multisession Radiosurgery (Experimental): Multisession Radiosurgery
  Interventions: Radiation: Multisession Radiosurgery

INTERVENTIONS:
Radiation: Multisession Radiosurgery — Patients will undergo multisession radiosurgery as clinical practice.
  Other Names: Cyberknife (Accuray)

SUMMARY:
Traditional treatment options for optic nerve sheath meningiomas (ONSM) include observation, surgery and radiotherapy, but to date none of these has become the clear treatment of choice.

The role of the radiotherapy remained uncertain because of the concern about radiation related optic neuropathy In the recent past two large series of patients treated with a fractionated stereotactic radiotherapy confirmed these positive experiences in tumour control and greatly reduced the concern about the treatment related toxicity.

Under the light of successful meningiomas treatment, radiosurgery, had proposed as a treatment option. Single session, high conformality, frame based radiosurgery systems are seldom if ever proposed as ONSMs treatment due to the known dose tolerance of the optic nerve.

The first experience in ONSMs treatment with multisession radiosurgery treatment was quite promising.

The aim of the present study is to prospectively evaluate the efficacy and safety of multisession radiosurgery in ONSMs treatment.

In order to evaluate multisession radiosurgery 50 patients will be enrolled in the present study.

All patients will be treated by using multisession radiosurgery, with 5 fractions of 5 Gy each to a total dose of 25 Gy prescribed to the 75-85% isodose line. Patients were evaluated both for tumor growth control and visual function.

DETAILED DESCRIPTION:
Introduction Optic Nerve Sheath Meningiomas (ONSMs) are rare tumours. They represent approximately the 2% of all orbital tumours, 1-2% of intracranial meningiomas and one third of the optic nerve lesions (23, 32, 42, 43). Usually these tumour are monolateral but 5% have a bilateral development (33) On the base of the growth pattern these tumours can be classified in primary and secondary forms. The former type arise from the arachnoid cap cell of the fibrous dural capsule of the optic nerve and they usually growth circumferentially along the nerve. Primary ONSMs can be further subdivided in orbital and intracanalicular forms.

Secondary ONSMs usually arise from the sphenoid ridge or the tuberculum sellae and subsequently spread into the optic canal and the orbit (14, 42).

Often the pathological studies show meningotheliomatous or transitional histology.

Middle aged woman are the most often affected (4, 36, 44). The most frequent presentation symptom is a visual loss, both in acuity or visual field. This is nearly an expression of an optic nerve direct compression and of the vascular rearrangement.

Optic nerve atrophy is common. Optociliary shunts are a late and rare sign but they are the direct expression of compressive optic neuropathy and it can be pathognomonic for the diagnosis of ONSM (35, 43).

Traditionally treatment options include observation, surgery and radiotherapy but, until now, any of these had assumed as the treatment of choice.

Nevertheless, the development of the new technology improved the interest in radiotherapy application.

Conservative treatment can be considered due to the benign nature of the meningiomas and their slow growth pattern. Nevertheless this unavoidably leads to a visual deterioration or complete blindness (18, 33, 43, 44).

Surgery is advocate for tumour administration, particularly in case of a progressive visual loss or complete blindness, tumour progression and intracranial involvement. Anyway because of their intimate relationship to the optic nerve, ophthalmic artery and central retina artery ONSMs complete removal is extremely challenging. Moreover post-operative course is often characterized by symptoms worsening (4, 8, 9, 15).

In the recent past, the role of the radiotherapy remained uncertain: many author reported a positive experience, but the concern about complication and secondary effects strongly limited its acceptance (4, 5, 16, 21, 22, 26, 29, 31, 32). Radiation optic neuropathy has been described following conventional radiotherapy treatments (45 Gy, 2 Gy per fraction) (40).

More recently two large series of patients treated with a fractionated stereotactic radiotherapy confirmed these positive experiences in tumour control and greatly reduced the concern about the treatment related toxicity (6, 27).

Under the light of successful meningiomas treatment, radiosurgery had proposed as a treatment option. Single session, high conformality, frame based radiosurgery systems are seldom if ever proposed as ONSMs treatment due to the known dose tolerance of the optic nerve (22).

The development of the radiosurgery technology, starting in 1994, introduced a new and effective therapeutic option (3, 11, 12).

In this way it is possible to exploit the different recovery speed of normal and pathological tissues to optimize the tumour control and at the same time to spare the surrounding structure avoiding damage to the visual pathways.

In fact, the comparison between various fractionation regimens resulting in roughly equivalent biologically equivalent dose (BED) for tumour control and normal tissue late effects (assuming that tumour and normal tissue late effect have a similar α/β ratio). In this way the acute (early) reactions would be reduced with larger fractions size (19).

The first experience in ONSMs treatment with multisession radiosurgery treatment was quite promising (32).

The aim of the present study is to prospectively evaluate the efficacy and safety of multisession radiosurgery in ONSMs treatment.

The treatment will be evaluated both in terms of tumour growth control and sparing for vision.

PATIENTS AND METHODS Patient's population. XX patients affected by an Optic Nerve Sheath Meningioma (ONSM), both orbital and intra-canalicular will be considered for a multisession radiosurgery.

Eligibility:

Inclusions criteria are a significant visual impairment at presentation, progression of visual dysfunction during the observation period, disease progression.

Due to the histological diagnosis imply an invasive and hazardous procedure, no biopsies will be performed and the diagnosis will be exclusively radiological.

Pre-treatment evaluation. All patients, before treatment, will be collectively evaluated by Neurosurgeon, Radiation Oncologist and Neuro-Ophthalmologist.

Clinical investigation includes a full neurological examination. Particularly the I, III, IV, V and VI pair of cranial nerve will be investigated.

Visual acuity, visual field will be also investigated by the same Neuro-ophthalmologist. Visual acuity will be investigated using best correct Snellen visual acuity. A standardized automated perimetry by humphrey Visual 30-2 field testing will be performed in order to define the presence of visual field deficits Dose selection and radiobiology considerations. The dose selection is based on previous experience with Radiosurgery and Stereotactical Radiotherapy (1, 2, 23, 28, 30), but also on the previous studies concerning the dose tolerance of the anterior visual pathways (38).

Assumed these considerations we plan multisession radiosurgery: all patients will be treated with a maximum dose of 25 Gy (5 Gy/fraction; 5 fractions).

The total dose plans in this study is comparable to the doses delivered with the conventional fractionated regimens (50,4 - 56 Gy). In fact, assumed that the meningioma's α/β ratio is approximately 3,7-3,8 Gy (34, 41).

According to the equivalent dose formula:

EQD2 = D * [(d + α/β)/(2 + α/β) = 38,2 Gy where D is the altered schedule total dose, d is the altered daily dose. Then, considering the differences between the overall treatment time between conventional fractionated and hypofractionated treatment (28 fractions, 5 fractions per week, 38 total days and 5 fractions, 5 days respectively), assumed Dprolif = 0,7 as for the most of the tumours (7, 17), where Dprolif is the dose recovered daily owning to proliferation: EQD2,T = EQD2,t - [(T - t) * Dprolif ] = 61 Gy Treatment planning. Patients will have a 1.25 mm thickness MRI, including fat suppression sequence, T1with Gadolinium sequence and a contrast-enhanced CT scans. The images will then merged in order to optimize the definition of the target volume and the intra-extraorbital segment of the optic nerve, and the organ at risk (i.e. retina) An inverse planning software will be adopted to optimize the target coverage and at the same time to achieve the maximum of conformality and homogeneity of the prescription dose. The treatment plan used for each treatment will be based on an analysis of the volumetric dose including dose-volume histogram (DVH) analyses of the PTV and critical normal structures. The number of paths and beams used for each patient will vary and will be determined by the selected individual treatment plan.

Target Volumes The target volume will consist of the tumor outlined in the treatment planning software seen on planning CT and/or MRI.

The planning target volume (PTV) is planned to encompasses the 75-85% isodose line. All organs at risk will be defined.

Follow-up. Following multisession radiosurgery, patients will be evaluated for tumour progression and visual function by a multidisciplinary team (Radiation Oncologist, Neurosurgeon; Neuro-Ophthalmologist). The patients will be evaluated 3 months after treatment, every 6 months during the first two years and then once per years.

Every follow-up includes Neurological, Radiological and neuro-ophthalmological evaluation.

Neuro-Ophthalmologic assessment includes a comprehensive evaluation of the visual acuity, visual field, extrinsic eyes movements, and proptosis. Visual acuity will be investigated by using the same tests at base line.

Post-treatment radiographic evaluation includes an MRI scan every 6 months. Primary end point Primary end points are local growth control and maintenance or improvement of visual acuity at base line Response criteria The partial response is defined as a tumour reduction more than 20 %. Progression disease is defined as any increase in the tumour dimensions.

Toxicity Ocular toxicity will be described with reference to CTCAE 3 version criteria. DATA COLLECTION Patients will be allocated a number and their data will be collected on a Case Report Forms. Data will include information from each protocol visit and will be completed on a timely manner.

STATISTICAL CONSIDERATIONS Analysis will be conducted to check if tumor control is correlated to clinical symptoms improvement by using short course radiotherapy treatment in relation to previous described radiobiological considerations.

Clinical improvement will be measured specific ophthalmological tests.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years old
* Patients with suspected optic nerve sheath meningioma (single lesion) Pain and/or neurologic deficit
* KPS ≥ 70
* Written consent

Exclusion Criteria:

* Pregnancy
* Bilateral meningioma or chiasma involved
* Allergy to contrast medium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
visual function outcome | 5 year
  pre and post treatment visual acuity and visual field will be evaluated

SECONDARY OUTCOMES:
PFS - progression free survival | 5 year
  Partial response: tumor reduction more than 20%. Progression disease: any increased
Safety: level of toxicity | 5 year
  Toxicity evaluated according to NCI CTCAE v3.0

CONTACTS AND LOCATIONS:
Overall Officials: Laura Fariselli, MD, Principal Investigator — Instittuto Nazionale Neurologico Carlo Besta
Locations (1):
- Instittuto Nazionale Neurologico Carlo Besta, Milan, Mi, Italy